CLINICAL TRIAL: NCT04870606
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Proxalutamide (GT0918) in Outpatients With Mild to Moderate COVID-19 Illness
Brief Title: Proxalutamide (GT0918) Treatment for Outpatients With Mild or Moderate COVID-19 Illness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GT0918-US-3001
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Efficacy and Safety
MeSH Terms: interventions — proxalutamide; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GT0918+ standard of care (Active Comparator): Proxalutamide 200mg, oral, QD, for continuous 14 days, plus standard of care(n=334)
  Interventions: Drug: Proxalutamide (GT0918)
- placebo+ standard of care (Placebo Comparator): Placebo 200mg, oral, QD, for continuous 14 days, plus standard of care(n=334)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proxalutamide (GT0918) — Proxalutamide (GT0918)+Standard of care determined by PI and local regulatory
  Other Names: standard of care
  Arms: GT0918+ standard of care
Drug: Placebo — Placebo+Standard of care determined by PI and local regulatory
  Other Names: standard of care
  Arms: placebo+ standard of care

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Proxalutamide (GT0918) as a treatment for outpatients COVID-19 subjects.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, multicenter study to evaluate the safety and efficacy of Proxalutamide (GT0918) in adult outpatients diagnosed with mild to moderate COVID-19. The study will be 2-arm comparison against matched placebo. The study will be conducted in around 100 sites in the USA and other countries. This study utilizes an adaptive design that maximizes our efficiency in identifying a safe and efficacious therapeutic agent for COVID-19 during the current outbreak. There will be an interim analysis after 334 subjects complete Day 28 after the first dose to allow early stopping for futility, efficacy, or safety. The study population will be subjects with mild to moderate COVID-19 illness chosen to evaluate if early intervention with anti-androgen therapy prior to respiratory compromise can effectively prevent progression to the severe form of COVID-19 illness. Randomization is essential for establishing efficacy of these new therapeutic agents.

The blood samples for PK analysis need to be collected for at least 200 subjects, whom will also be randomized into the interventional treatment or placebo group with 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legally authorized representative give signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
2. Understand and agree to comply with planned study procedures.
3. Male subjects with age ≥18 years of age at the time of randomization.
4. Are currently not hospitalized.
5. Have one or more mild or moderate symptom(s) COVID-19-related symptoms within 5 days of onset of symptoms onset
6. Must have first positive SARS-CoV-2 viral infection determination (has laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen) ≤3 days prior to start of the first dose.
7. Regardless of their fertility status, male subjects must agree to either remain abstinent (if this is their preferred and usual lifestyle) or use condoms as well as one additional highly effective method of contraception (less than 1% failure rate) or effective method of contraception with nonpregnant women of childbearing potential partners for the duration of the study and until 90 days after the last dose.

   Use an acceptable method of contraception such as:
   * Highly effective methods of contraception (less than 1% failure rate) comprise, but are not limited to

     * combination oral contraceptives
     * implanted contraceptives, or
     * intrauterine devices.
   * Effective methods of contraception comprise but are not limited to

     * diaphragms with spermicide or cervical sponges.
     * men and their partners may choose to use a double-barrier method of contraception that must include use of a spermicide.
8. Agree to the collection of nasopharyngeal swabs and venous blood.

Exclusion Criteria:

1. Have SpO2 ≤ 93% on room air at sea level or PaO2/FiO2 < 300, respiratory rate ≥30 per minute, heart rate ≥125 per minute
2. Estimated glomerular filtration rate (eGFR) < 30 ml/min
3. Serum total bilirubin > 1.5 x ULN (upper limit of normal) and AST and ALT >3x ULN
4. Subjects with significant cardiovascular disease as following:

   i. heart failure NYHA class ≥3 ii. left ventricular ejection fraction <50% iii. those with a history of cardiac arrhythmias, including long QT syndrome.
5. Has been admitted to a hospital prior to randomization, or is hospitalized (inpatient) at randomization, due to COVID-19 or requires treatment with supplemental oxygen.
6. Have known allergies to any of the components used in the formulation of the interventions.
7. Have hemodynamic instability requiring use of vasopressors within 24 hours of randomization.
8. Suspected or proven serious, active bacterial, fungal, viral, or other infection (except COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention (i.e. known history of human immunodeficiency virus [HIV]).
9. Have any co-morbidity requiring surgery within <7 days, or that is considered life-threatening within 30 days.
10. Have any serious concomitant systemic disease, condition, or disorder that, in the opinion of the investigator, should preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 733 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Lu, Study Director — Suzhou Kintor Pharmaceuticals,Inc.
Locations (8):
- United States (8):
  - Absolute Clinical Research, Phoenix, Arizona
  - Long Beach Clinical Trials, Long Beach, California
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Olivo Medical and Wellness Center, Chicago, Illinois
  - Gtc Research, Shawnee Mission, Kansas
  - Platinum Research Network, LLC, Metairie, Louisiana
  - Main Street Physician's Care, Little River, South Carolina
  - Lotus Clinical Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 865 subjects were screened, of whom 132 subjects failed at screening. A total of 733 subjects were randomized in this study
Pre-assignment Details: 733 subjects were randomized. 366 subjects were assigned to receive Pruxelutamide arm and 367 subjects were assigned to receive placebo arm. All randomized subjects were included in the ITT population.
  730 subjects, which included 365 subjects from each of the Pruxelutamide and placebo groups, were randomized and received at least one dose of treatment. These subjects were included in both the mITT and SS populations.
Period: Overall Study
Arm/Group | GT0918+ Standard of Care | Placebo+ Standard of Care
Started | 366 | 367
Received at Least One Dose of Treatment After Randomised | 365 | 365
Completed | 354 | 359
Not Completed | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GT0918+ Standard of Care | Placebo+ Standard of Care | Total
Number analyzed (Participants) | 366 | 367 | 733
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (13.82) | 40.9 (13.45) | 41 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 185 | 368
  Male | 183 | 182 | 365
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 322 | 325 | 647
  Not Hispanic or Latino | 44 | 42 | 86
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 25 | 33 | 58
  White | 323 | 316 | 639
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 13 | 29
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.02 (5.817) | 29.03 (6.625) | 29.02 (6.040)
Vaccination Status [Count of Participants; unit: Participants]
  Fully Vaccinated | 140 | 152 | 292
  Partially Vaccinated | 14 | 16 | 30
  Non Vaccinated | 210 | 194 | 404
  Unknown | 2 | 5 | 7
COVID-19 Test Type [Count of Participants; unit: Participants]
  Molecular (RNA or PCR) Test | 228 | 236 | 464
  Antigen (Rapid) Test | 137 | 127 | 264
  Unknown | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Efficacy in Terms of Clinical Status Following Treatment With Pruxelutamide (GT0918) Compared to Placebo
Description: In mITT (administrated at least one dose)，percentage of subjects who do not experience any of the following events due to all causes by Day 28:
  * Hospitalization for ≥ 24 hours, or
  * Supplemental oxygen for ≥24 hours in response to SpO2 ≤93%, or
  * Death
Time Frame: 28 days
Population: In mITT (administrated at least one dose)
Measure: Count of Participants; unit: Participants
Arm/Group | GT0918+ Standard of Care | Placebo+ Standard of Care
Number analyzed (Participants) | 365 | 365
Participants | 361 | 357

2. Primary Outcome: Sensitivity Analysis to Evaluate Efficacy in Terms of Clinical Status Following Treatment With Pruxelutamide (GT0918) Compared to Placebo
Description: In mITT (treatment period >7 days) , percentage of subjects who do not experience any of the following events due to all causes by Day 28:
  * Hospitalization for ≥ 24 hours, or
  * Supplemental oxygen for ≥24 hours in response to SpO2 ≤93%, or
  * Death
Time Frame: 28 days
Population: mITT (treatment period >7 days) The mITT was defined as patients treated at least one dose. The primary outcome was analyzed based on mITT set.
  At the same time, the sponsor did some sensitive analysis based on another mITT set, defined as patients treated longer than 7 days, to support the primary outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | GT0918+ Standard of Care | Placebo+ Standard of Care
Number analyzed (Participants) | 348 | 345
Participants | 348 | 339
Statistical Analysis 1: Comparison: GT0918+ Standard of Care vs Placebo+ Standard of Care; Test type: Superiority; p = 0.0181, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 0.025

3. Secondary Outcome: Proportion of Subjects With Hospitalization by Day 28
Description: Percentage of subjects who do experience any of the following events due to all causes by Day 28:
  * Hospitalization for ≥ 24 hours, or
  * Supplemental oxygen for ≥24 hours in response to SpO2 ≤93%, or
  * Death
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | GT0918+ Standard of Care | Placebo+ Standard of Care
Number analyzed (Participants) | 365 | 365
Participants | 4 | 8
Statistical Analysis 1: Comparison: GT0918+ Standard of Care vs Placebo+ Standard of Care; Test type: Superiority; p = 0.1223, Chi-squared; Mean Difference (Final Values) = 0.025

4. Secondary Outcome: Viral Load
Description: Changes from baseline in SARS-CoV-2 viral load at days 3, 7, 14, and 28.
Time Frame: at day 3,7,14,28
Population: The patient enrolled by local laboratory-confirmed SARS-CoV-2 infection; at the same time, Quantitative RT-qPCR done in the central laboratory was to determine the viral load change from different time points." Only the patients with positive dd-PCR test results, Limit of Detection with 59.9 copies/mL, were included in the viral load analysis, 277 patients in GT0918 group and 272 patients in placebo group.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | GT0918+ Standard of Care | Placebo+ Standard of Care
Number analyzed (Participants) | 277 | 272
log10 copies/mL
  Days28 | -5.4 (0.1) | -4.9 (0.1)
  Days14 | -4.8 (0.11) | -4.5 (0.12)
  Days 7 | -3.6 (0.12) | -3.4 (0.13)
  Days 3 | -2.0 (0.12) | -1.5 (0.12)
Statistical Analysis 1: Comparison: GT0918+ Standard of Care vs Placebo+ Standard of Care; Test type: Superiority; p = 0.0038, t-test, 2 sided; Mean Difference (Final Values) = 0.025

ADVERSE EVENTS:
Time Frame: Up to day 42; the investigator (and/or designee) documented all AEs reported by the subject from the time subjects given consent through completion of the EOS visit (day42) per protocol
Description: If an event is not an AE per definition, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under study, death due to progression of disease).
  Hospitalizations related to routine treatment or monitoring of the studied indication, not associated with any deterioration in condition should not be reported as SAEs.
Arm/Group | GT0918+ Standard of Care | Placebo+ Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/365 | 1/365
Serious Adverse Events (participants affected / at risk) | 0/365 | 0/365
Other Adverse Events (participants affected / at risk) | 19/365 | 11/365
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GT0918+ Standard of Care (N=365) | Placebo+ Standard of Care (N=365)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0)
Vertigo (Nervous system disorders) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2)
Fibrin D dimer increased (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04870606/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT04870606/SAP_001.pdf
  • Informed Consent Form (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT04870606/ICF_002.pdf